CLINICAL TRIAL: NCT00016965
Title: A Phase II Trial of Epothilone B Analogue BMS-247550 (NSC #710428) Every 21 Days in Patients With Advanced Pancreas Cancer
Brief Title: BMS-247550 in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068636; SWOG-S0107
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2003-04

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ixabepilone

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BMS-247550 in treating patients who have advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 6-month survival rate and time to treatment failure in patients with advanced pancreatic adenocarcinoma treated with BMS-247550.
* Determine the frequency and severity of toxic effects of this drug in these patients.
* Determine the complete and partial response in those patients with measurable disease treated with this drug.
* Determine the pharmacokinetic profile of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive BMS-247550 IV over 3 hours on day 1. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression.

Patients are followed every 6 months for 2 years and then annually until 3 years after registration.

PROJECTED ACCRUAL: A total of 25-55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced pancreatic adenocarcinoma

  * Distant metastases OR
  * Locoregional disease that has failed or is not amenable to locoregional therapy
* No de novo locoregional disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* Adult

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2.5 times ULN
* Alkaline phosphatase less than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No recent myocardial infarction, unstable angina, or life-threatening arrhythmia

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I or II cancer in remission
* No prior severe hypersensitivity reaction to drugs containing Cremophor EL
* No active or uncontrolled infection
* No severe psychiatric disorders

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior neoadjuvant, adjuvant, or primary immunotherapy for advanced pancreatic cancer
* No concurrent anticancer immunotherapy

Chemotherapy:

* No prior neoadjuvant, adjuvant, or primary chemotherapy for advanced pancreatic cancer
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* No prior neoadjuvant, adjuvant, or primary hormonal therapy for advanced pancreatic cancer
* No concurrent anticancer hormonal therapy

Radiotherapy:

* No prior neoadjuvant, adjuvant, or primary radiotherapy or chemoradiotherapy for advanced pancreatic cancer
* Prior palliative radiotherapy allowed if at least 1 lesion remains outside of radiation field or at least 1 lesion has progressed since radiotherapy
* No concurrent anticancer radiotherapy except palliative radiotherapy to non-target metastatic sites

Surgery:

* At least 2 weeks since prior surgery for pancreatic cancer and recovered

Other:

* No other concurrent anticancer therapy
* No concurrent herbal or unconventional therapy (e.g., St. John's Wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Whitehead, MD, Study Chair — University of Texas
Locations (95):
- United States (95):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Genesis Medical Center, Davenport, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Oregon Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Whitehead RP, McCoy S, Rivkin SE, Gross HM, Conrad ME, Doolittle GC, Wolff RA, Goodwin JW, Dakhil SR, Abbruzzese JL. A Phase II trial of epothilone B analogue BMS-247550 (NSC #710428) ixabepilone, in patients with advanced pancreas cancer: a Southwest Oncology Group study. Invest New Drugs. 2006 Nov;24(6):515-20. doi: 10.1007/s10637-006-8440-x. PMID 16699973